CLINICAL TRIAL: NCT01907022
Title: Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) in Combination With Relaxation Therapy in Patients With Chronic Tinnitus
Brief Title: Combined rTMS and Relaxation in Chronic Tinnitus
Acronym: RELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, PhD, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Reg-Ti-CDC01-RELAX
Record Dates: First submitted 2013-07-19; First posted 2013-07-24 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Tinnitus
Keywords: repetitive transcranial magnetic stimulation; chronic tinnitus; relaxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Left dorsolateral prefrontal cortex (DLPFC) Butterfly Coil (Experimental): High frequency rTMS ( Alpine Biomed Mag Pro Option): 2000 stimuli of 20 Hz over the left DLPFC (each session), Butterfly-water-cooled-Coil, 110% motor threshold; followed by: low frequency rTMS ( Alpine Biomed Mag Pro Option) applied over left temporoparietal cortex, Butterfly-water-cooled-Coil (2000 Stimuli of 1 Hz each session), 110% motor threshold. Relaxation therapy during the 1Hz stimulation with external audio tape instructions.
  Interventions: Device: Left DLPFC Butterfly Coil

INTERVENTIONS:
Device: Left DLPFC Butterfly Coil — High frequency rTMS ( Alpine Biomed Mag Pro Option): 2000 stimuli of 20 Hz over the left DLPFC (each session), Butterfly-water-cooled-Coil, 110% motor threshold; followed by: low frequency rTMS ( Alpine Biomed Mag Pro Option) applied over left temporoparietal cortex, Butterfly-water-cooled-Coil (2000 Stimuli of 1 Hz each session), 110% motor threshold. Relaxation therapy during the 1Hz stimulation with external audio tape instructions.
  Arms: Left DLPFC Butterfly Coil

SUMMARY:
Repetitive Transcranial Magnetic Stimulation in combination with relaxation therapy is used to modulate the neural pathways contributing to the perception and distress of phantom sounds.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. One significant modulator of tinnitus is stress. Tinnitus has been shown to be generated in the brain, as a result of functional reorganization of auditory neural pathways and the central auditory system. Also non-auditory cortical areas of attention allocation and emotional processing was shown to be involved. Treatment remains difficult. The most effective treatment in chronic tinnitus is cognitive behavioral therapy including elements of relaxation therapy. Repetitive transcranial magnetic stimulation (rTMS) is also effective in treatment of tinnitus with moderate effect size. Pilot data were positive for low-frequency rTMS applied to the temporoparietal areas and high-frequency rTMS applied to the left frontal cortex. Newer findings indicate that exercise-combined non-invasive brain stimulation might show superior effects in contrast to rTMS or exercise alone. Combination of relaxation and two-sided (frontal and temporo-parietal) rTMS will be examined with regard to feasibility, safety and clinical efficacy in patients suffering from chronic tinnitus in a pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bothersome, subjective chronic tinnitus
* Duration of tinnitus more than 6 months

Exclusion Criteria:

* Objective tinnitus
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Prior treatment with TMS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of treatment responders (TQ reduction > 5, contrast Baseline versus end of treatment) | Week 12

SECONDARY OUTCOMES:
Change of tinnitus severity as measured by the Tinnitus Questionaire of Goebel&Hiller | Week 4
Change of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI) | Week 4
Change of tinnitus severity as measured by the Tinnitus Severity Scale | Week 4
Change of tinnitus severity as measured by the Tinnitus Questionaire of Goebel&Hiller | Week 2
Change of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI) | Week 2
Change of tinnitus severity as measured by the Tinnitus Severity Scale | Week 2
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Week 4
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Week 2
Change in quality of life as measured by the World Health Organization Quality of Life (WHOQoL) | Week 2
Change in quality of life as measured by the World Health Organization Quality of Life(WHOQoL) | Week 4
Change of tinnitus severity as measured by the Tinnitus Questionaire of Goebel&Hiller | Week 12
Change of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI) | Week 12
Change of tinnitus severity as measured by the Tinnitus Severity Scale | Week 12
Change in quality of life as measured by the World Health Organization Quality of Life (WHOQoL) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Ph.D., Principal Investigator — University of Regensburg - Dept of Psychiatry
Locations (1):
- University of Regensburg - Dept of Psychiatry, Regensburg, Germany